CLINICAL TRIAL: NCT04897191
Title: Assessing Age-dependent Reference Values for Microvascular Structure and Function in Healthy Participant Together With Macrovascular Function With Optical Coherence Tomography Angiography
Brief Title: Healthy Age-dependent Reference Values for Microvascular Structure and Function
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Surrey (Other)
Responsible Party: Sponsor
Other Study IDs: OCTA1
Record Dates: First submitted 2021-05-18; First posted 2021-05-21 (Actual); Last update posted 2021-05-21 (Actual); Status verified 2021-05

CONDITIONS: Vascular Endothelium; Microvascular Circulation; Arterial Stiffness; Healthy Ageing
MeSH Terms: interventions — Aging

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Healthy: Healthy people age 20-70 years
  Interventions: Other: Age

INTERVENTIONS:
Other: Age — Determination of age-dependence

SUMMARY:
The greatest challenge in our ageing society are cardiovascular diseases such as stroke, heart attack, peripheral artery disease of the legs with non-healing wounds (ulcers), or diabetes. How healthy ageing affects the smallest blood vessels (microcirculation) and is not well understood. One reason for this is that no generally available medical instrument has the resolution to study the microcirculation. The recently developed optical coherence tomography angiography (OCTA), currently mainly used by eye doctors, is able to visualise the microcirculation. We have developed an automated software (OCTAVA) to determine metrics to characterise the microcirculation on the layers of density, diameter and tortuosity.

In the current study we aim at providing reference values of these metrics in hands and feet of healthy people according to age together with macrovascular function in arms and legs.

ELIGIBILITY:
Inclusion criteria:

Healthy, 20-70 years, BMI 20-30 kg/m^2

Exclusion criteria:

Diabetes mellitus, symptoms of acute infection, cardiac arrhythmias, active malignancy, clinical signs or symptoms of cardiovascular disease (coronary artery disease, lower extremity artery disease, cerebrovascular disease): angina pectoris, dyspnea, palpitation, syncope, claudication, active vasoactive medication.

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthy adults aiming at n=10 of each decade
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2021-05-18 (Actual); Primary Completion 2021-07 (Estimated); Study Completion 2021-08 (Estimated)

PRIMARY OUTCOMES:
Microvascular density | 1 day (One timepoint during single visit)
  Density of skin microvasculature of hand and foot with OCTA at rest and after 5 min distal occlusion
Microvascular diameter | 1 day (One timepoint during single visit)
  Diameter of skin microvasculature of hand and foot with OCTA at rest and after 5 min distal occlusion
Microvascular turtuosity | 1 day (One timepoint during single visit)
  Turtuosity of skin microvasculature of hand and foot with OCTA at rest and after 5 min distal occlusion

SECONDARY OUTCOMES:
Blood pressure | 1 day (One timepoint during single visit)
  Upper arm blood pressure and leg systolic blood pressure
Endothelial function | 1 day (One timepoint during single visit)
  Flow-mediated dilation of brachial and common femoral artery with ultrasound
Arterial stiffness | 1 day (One timepoint during single visit)
  Pulse wave velocity measured at upper arm (Arteriograph)
Arterial stiffness | 1 day (One timepoint during single visit)
  Pulse wave velocity measured with photoplethysmography sensors at hand and foot

CONTACTS AND LOCATIONS:
Overall Officials: Christian Heiss, Prof., Principal Investigator — University of Surrey
Locations (1):
- University of Surrey, Guildford, United Kingdom

IPD SHARING:
Plan to Share IPD: No
Depending on outcome, we may publish IPD.